CLINICAL TRIAL: NCT06137846
Title: Treatment of Peri-implant Mucositis and Supportive Peri-implant Therapy Using an Erythritol Air- Polishing Device Versus Conventional Mechanical Debridement: A 6-month Randomized Controlled Clinical Trial
Brief Title: Treatment of Peri-implant Mucositis and Supportive Peri-implant Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Hom-Lay Wang, DDS, MSD, Ph D, Collegiate Professor of Periodontics and Professor of Dentistry, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00164918
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Peri-implant Mucositis
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Peri-mucositis (Experimental): Dental implant has peri-implant mucositis
  Interventions: Device: Air-Polish; Device: Ultrasonic
- Healthy (Placebo Comparator): Dental implant does not have peri-implant mucositis
  Interventions: Device: Air-Polish

INTERVENTIONS:
Device: Air-Polish — Dental implant will be cleaned with an airpolishing device
Device: Ultrasonic — Dental implant will be cleaned with an ultrasonic device with a plastic tip
  Arms: Peri-mucositis

SUMMARY:
The investigators are evaluating the therapeutic outcomes of two cleaning instruments on treating peri-implant mucositis. Peri-implant mucositis is inflammation around an implant that is limited to only the gum tissue and is characterized by bleeding on probing, pus, and without any evidence of bone loss. The investigators wish to compare the amount of inflammation and bacteria through measurements (like probing depth) and by collecting fluid and plaque samples around participants' implant after using one of the two cleaning instruments.

DETAILED DESCRIPTION:
Despite the potential benefits of an air-polishing device with erythritol powder, clinical trials using the device as a monotherapy for treating patients with peri-implant mucositis remained limited. Therefore, the primary aim of the present study is to compare clinical outcomes of the non-surgical treatment of peri-implant mucositis and subsequent supportive peri-implant therapy (SPIT) using an erythritol air-polishing device or conventional mechanical debridement. The secondary aim is to compare the resolution of inflammation after non-surgical treatment of peri-implant mucositis and to monitor levels of peri-implant tissues inflammation during supportive peri-implant therapy by using the level of selected pro-inflammatory cytokines.

Up to 60 participants with dental implants will be recruited from patients seeking and/or receiving dental care at the University of Michigan Graduate Periodontics department, until 34 peri-mucositis participants and 17 healthy participants are achieved.

ELIGIBILITY:
Inclusion criteria:

1. Age 18 to 85 years.
2. Healthy systemic conditions (American Society of Anesthesiologists classification (ASA) I or II: systemically healthy or suffer from mild to moderate, but well controlled systemic diseases).
3. Must have at least one osseointegrated dental implant with the following conditions (Berglundh et al. 2018a).

   * At least 12 months since the prosthesis was placed.
   * Absence of bone loss beyond crestal bone level changes from initial bone remodeling.
   * For implant mucositis subjects: Presence of bleeding and/or suppuration on gentle probing around implant at least 2 sites. Visual inspection demonstrating the presence of peri-implant signs of inflammation.
   * For healthy implant subjects: Absence of bleeding and/or suppuration on gentle probing around implant.
4. Have a current (less than 6 months old) x-ray of the affected site
5. All participants must be enrolled in a 3 to 6 months maintenance recall program including teeth/implants prophylaxis and supportive periodontal therapy.

Exclusion criteria:

1. Poorly controlled diabetes mellitus (HbA1c >6.5).
2. Uncontrolled systemic disease or condition known to alter bone metabolism. (e.g. osteoporosis, osteopenia, hyperparathyroidism, Paget's disease)
3. Current smokers or vapers.
4. Pregnancy or could be pregnant (self-reported), or plan to be pregnant in the next 6 months.
5. Long-term (3 months) intake of anti-inflammatory medications (e.g. non-steroidal anti-inflammatory drugs (NSAIDs)) known to affect periodontal status within one month previous to participation in the study.
6. Taking corticosteroids.
7. Long-term antibiotic use (> one weeks) within three months previous to participation in the study.
8. No history of supragingival scaling or non-surgical therapy at the affected implant site in the last 1 month.
9. Taking anticoagulant medications.
10. Subjects who require prophylactic antibiotics.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2023-10-31 (Actual); Primary Completion 2025-03-19 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
Probing depth measurements | Baseline, 2 weeks, 4 weeks, 3 months, and 6 months
  To compare probing depth measurements in millimeters after non-surgical treatment of peri-implant mucositis
Bleeding on probing scores (Mombelli et al.) | Baseline, 2 weeks, 4 weeks, 3 months, and 6 months
  To compare bleeding on probing after non-surgical treatment of peri-implant mucositis. Possible scores range from 0 to 3, with higher scores indicating heavier bleeding.
Plaque score (Loe & Silness) | Baseline, 2 weeks, 4 weeks, 3 months, and 6 months
  To compare plaque scores after non-surgical treatment of peri-implant mucositis. Possible scores range from 0 to 3, with higher scores indicating greater plaque accumulation.
Gingival index (Loe & Silness) | Baseline, 2 weeks, 4 weeks, 3 months, and 6 months
  To compare gingival index scores after non-surgical treatment of peri-implant mucositis. Possible scores range from 0 to 3, with higher scores indicating greater inflammation.
Gum recession measurement | Baseline, 2 weeks, 4 weeks, 3 months, and 6 months
  To compare gum recession after non-surgical treatment of peri-implant mucositis
Bone measurement | Baseline, 3 months, and 6 months
  Loss of supporting bone measured by standardized radiographs

SECONDARY OUTCOMES:
Inflammatory cytokines levels | Baseline, 2 weeks, 4 weeks, 3 months, and 6 months
  To compare changes in the level of inflammatory cytokines in peri-implant crevicular fluid (PICF)
Bacterial DNA levels | Baseline, 2 weeks, 4 weeks, 3 months, and 6 months
  To compare changes in the level of bacterial DNA of Aa, Pg, Pi, Tf, and Td in PICF

CONTACTS AND LOCATIONS:
Overall Officials: Hom-Lay Wang, DDS MSD PhD, Principal Investigator — Department of Periodontics and Oral Medicine University of Michigan
Locations (1):
- University of Michigan School of Dentistry, Ann Arbor, Michigan, United States